CLINICAL TRIAL: NCT00124761
Title: A Randomised Trial of Surgery Plus Whole Brain Radiotherapy (WBRT) Versus Radiosurgery Plus WBRT for Solitary Brain Metastases
Brief Title: A Trial Comparing Radiosurgery With Surgery for Solitary Brain Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Adelaide Hospital (Other)
Responsible Party: A/Prof Daniel Roos, Royal Adelaide Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021108
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Neoplasm Metastasis; Brain Neoplasm
Keywords: Radiosurgery; Brain metastases; Whole Brain Radiotherapy; Neurosurgery; Solitary Brain Metastases; Adult Tumours Metastatic to Brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Surgical Procedures, Operative; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery + Whole Brain Radiotherapy (Other)
  Interventions: Procedure: Surgery + WBRT
- RadioSurgery + Whole Brain Radiotherapy (Experimental)
  Interventions: Radiation: Radiosurgery + WBRT

INTERVENTIONS:
Procedure: Surgery + WBRT — Surgery - complete excision of Solitary Brain Metastasis with 30 Gy in 10 fractions over 2 2 1/2 weeks
  Other Names: S + WBRT
  Arms: Surgery + Whole Brain Radiotherapy
Radiation: Radiosurgery + WBRT — Radiosurgery - Marginal dose based on maximum tumour diameter
  Other Names: RS + WBRT
  Arms: RadioSurgery + Whole Brain Radiotherapy

SUMMARY:
This study examines surgery versus radiosurgery (highly focussed radiation) for the treatment of cancer which has spread to one spot in the brain (solitary brain "metastasis"). For these two treatment options, it will compare patients' survival times, quality of life, control rate of the brain metastases and side effects. It uses the most rigorous scientific method available called "randomisation" which minimises biases that exist with other types of studies. It will involve 30 - 40 patients.

DETAILED DESCRIPTION:
Primary objectives - to evaluate for solitary brain metastases whether both overall survival and health related quality of life (HQoL) in patients treated with radiosurgery (RS) plus whole brain radiotherapy (WBRT) are non-inferior to those of patients treated with surgery (S) plus WBRT.

Secondary objectives - to compare between the two treatment arms time to local and distant brain recurrence, failure free survival, acute and late toxicity.

Hypothesis - Patients treated with RS + WBRT have neither worse survival nor worse quality of life than those treated with S + WBRT.

Research plan:

* Trial design - Single-centre prospective randomised Phase III controlled two arm non-inferiority study with the "gold standard" of surgery (plus WBRT) as the control arm. Blinding to trial arm will not be feasible. Stratification is by Radiation Therapy Oncology Group Recursive Partitioning Analysis (RPA) prognostic Class 1 vs 2 vs 3.
* Main eligibility criteria - single presumed metastasis on MRI brain; systemic cancer diagnosed within the last 5 years; considered suitable for both S and RS; written informed consent.
* Main exclusion criteria - surgery indicated for life-threatening raised intra-cranial pressure or tissue diagnosis; surgery contra-indicated by site or medical co-morbidities; leptomeningeal disease; primary is small cell lung cancer, germ cell tumour, lymphoma, leukaemia or myeloma.
* Radiation - WBRT dose is 30 Gy in 10 fractions over 2 weeks. RS dose is based on lesion size up to 4 cm (15-20 Gy).
* Surgery - Aim is complete excision.
* Treatment sequence and patient assessments - Any sequencing of S/RS and WBRT is allowable, as long as the brain treatment is commenced within 2 weeks after, and completed within 6½ weeks after the diagnostic MRI brain. Assessments at baseline, during brain treatment, at 2 and 3 months after commencement, then 3 monthly, with MRI brain at 3 and 6 months, and/or as clinically indicated. Acute toxicity monitored by NCI Common Toxicity Criteria, late toxicity by RTOG/EORTC Late Radiation Morbidity Scheme. HQoL assessed by EORTC QLQ-C30 and QLQ-BN20.
* Sample size - 30-40 patients over 5 years.

Outcomes and Significance:

The trial will enable Level I evidence to be applied to this common clinical problem. Patients will be able to make an informed choice based upon valid survival, quality of life and toxicity comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Single presumed brain metastasis on contrast magnetic resonance imaging (MRI) scan within two weeks before commencement of treatment.
* Systemic cancer diagnosed histologically or cytologically synchronous with, or within 5 years of treatment of the presumed brain metastasis (other than non-melanoma skin cancer and cancer in-situ of the cervix, neither of which would be reasonably attributable as the primary site). Exception - melanoma diagnosed > 5 years previously is allowable in view of the extremely variable natural history of melanoma.
* Age >= 18 (no upper age limit).
* Considered suitable for both S and RS by the neurosurgeon and radiation oncologist (see exclusions).
* Patient must agree to adjuvant WBRT.
* RTOG RPA Class 1 or 2 (Karnofsky Performance Status [KPS] >= 70 after adequate trial of corticosteroids).
* RPA Class 3 patients (KPS < 70) eligible if it is considered that the poor performance status is due primarily to the solitary metastasis, aggressive local treatment of which may be expected to restore good performance status. This would ordinarily be associated with minimal systemic disease burden.
* Accessible for treatment and follow-up.
* Patient is infertile or is aware of the risk of becoming pregnant or fathering children and will use adequate contraception.
* Written informed consent

Exclusion Criteria:

* Previous history of brain metastasis(es)
* Surgery indicated to relieve life-threatening raised intracranial pressure or excision required for tissue diagnosis (no extra-cranial site to biopsy ie unknown primary). However, prior diagnostic (non-excisional) biopsy is allowable - it is acknowledged that the 50% probability of a repeat surgical procedure on subsequent randomisation would not be acceptable to many patients and clinicians.
* Surgery contraindicated by site (e.g. thalamus, brain stem) or medical co-morbidities.
* Leptomeningeal disease.
* Primary is small cell lung cancer, germ cell tumour, lymphoma, leukaemia or myeloma.
* Prior cranial RT (including RS).
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-12; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Overall survival and Quality of life | Until death or study completion

SECONDARY OUTCOMES:
Local and distant recurrence | Until death or study completion
Failure free survival | Until death or study completion
Acute and late toxicities | Acute toxicities 6 weeks post RT and late toxicities until death

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roos, MD, FRANZCR, Study Chair — Royal Adelaide Hospital
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Roos DE, Brophy BP, Zavgorodni SF, Katsilis ES. Radiosurgery for brain metastases at the Royal Adelaide Hospital: are we treating the right patients? Australas Radiol. 2002 Dec;46(4):402-8. doi: 10.1046/j.1440-1673.2002.t01-1-01094.x. PMID 12452912
- [Derived] Roos DE, Smith JG, Stephens SW. Radiosurgery versus surgery, both with adjuvant whole brain radiotherapy, for solitary brain metastases: a randomised controlled trial. Clin Oncol (R Coll Radiol). 2011 Nov;23(9):646-51. doi: 10.1016/j.clon.2011.04.009. Epub 2011 May 17. PMID 21592754